CLINICAL TRIAL: NCT06045351
Title: Efficacy of Vitamin D Supplementation in Females With Polycystic Ovary Syndrome: a Randomized Open Label Delayed-start Design
Brief Title: Efficacy of Injectable Vitamin D Supplementation in Females With Polycystic Ovary Syndrome
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Pakistan Science Foundation (Other)
Responsible Party: Principal Investigator, Rehana Rehman, Professor, Aga Khan University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AKUBBS
Record Dates: First submitted 2023-09-05; First posted 2023-09-21 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Anovulatory Infertility
Keywords: Poly cystic Ovarian Syndrome; randomized open label trial; delayed-start design; vitamin D; Pakistan
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: Infertile females with Polycystic Ovarian Syndrome
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VD supplementation (Experimental): Experimental Group (Group A; n=71):
  The intervention (experimental) group will receive VD injections 600,000 I.U I/M once with 1 gram calcium supplemental daily in the initial 12 weeks. After that standard PCOS care; i) Glucophage XR 750 mg (once for 15 days then twice daily) ii) progesterone supplementation (1 capsule Progeffik 100 mg every 3 weeks, then 1 week off) and iii) calcium supplements will be given for next 12 weeks.
  Interventions: Drug: Vitamin D
- Control (Active Comparator): Control Group (Group B; n=71):
  Participants will receive standard PCOS treatment; Glucophage XR 750 mg once at dinner for 15 days then twice daily and Capsule Progeffik 100 mg once at night every 3 weeks, then 1 week off for initial-- 12 weeks.
  Then VD supplementation (600,000 IUI/M) will be given once during the study period with Calcium 1000 mg/day and continued Standard PCOS treatment from 12- 24 weeks
  Interventions: Other: Active Comparator

INTERVENTIONS:
Drug: Vitamin D — Intervention Group Initial 12 weeks;
  * VD supplementation (600,000 IU I/M) once during the study period
  * Elemental calcium 1000 mg/day From 12-24 weeks: Standard PCOS;
  * Glucophage XR 750 mg once at dinner for 15 days then twice daily
  * Capsule Progeffik 100 mg once at night every 3 weeks, then 1 week off
  * Calcium 1000 mg/day
  Other Names: Experimental; Group A
  Arms: VD supplementation
Other: Active Comparator — Active Comparator (Group B; n=71):
  Initial-- 12 weeks;
  * Standard PCOS;
  * Glucophage XR 750 mg once at dinner for 15 days then twice daily
  * Capsule Progeffik 100 mg once at night every 3 weeks, then 1 week off From 12- 24 weeks
  * VD supplementation (600,000 IUI/M) once during the study period
  * Calcium 1000 mg/day
  * Standard PCOS Continued
  Other Names: Group B
  Arms: Control

SUMMARY:
Poly cystic Ovarian Syndrome (PCOS) is an endocrine disorder of reproductive age defined by "the presence of any two out of three criteria: oligo and/or anovulation, excess androgen activity and/or polycystic ovarian morphology on ultrasound". Considering role of vitamin D (VD) (3, 4) and high prevalence (58%) of deficiency in PCOS of Pakistan. Researchers hypothesized that its correction would improve response to standard PCOS treatment. The objective is to compare PCOS parameters in intervention group (Group A) receiving VD supplementation and then PCOS care with control group (Group B) receiving standard PCOS care and then VD supplementation. A randomized open label trial: delayed-start design will be conducted on VD deficient PCOS females VD < 20ng/ml ; Group A will receive VD injections 600,000 I.U I/M once with 1 gram calcium supplement daily in the initial 12 weeks. After that standard PCOS care; i) Glucophage XR 750 mg (once for 15 days then twice daily) ii) progesterone supplementation (1 capsule Progeffik 100 mg every 3 weeks, then 1 week off) and iii) calcium supplements will be given for next 12 weeks. PCOS females in Group B will receive standard PCOS care (same) with addition of VD and calcium supplementation after 12 weeks till study end point. Study outcomes will be comparison of i) hyperandrogenism by Free Androgen Index [Total Testosterone, Steroid Hormone Binding Globulin ii) insulin Resistance by HOMA-IR (serum Insulin, Fasting Blood Glucose) and iii) oxidative stress by Total Antioxidant Capacity after 24-weeks in these Groups'd levels after supplementation will be assessed for confirmation of correction and calcium and albumin levels for detection of hypercalcemia. Results of this study will inform the clinicians to add VD before or after the standard PCOS care for rectification of endocrine and metabolic derangements as a cost-effective treatment and prevention strategy in these females.

DETAILED DESCRIPTION:
This study will comprise of two groups (A and B) with 71 participants in each group carried for a duration of 24 weeks.

Intervention Details for Group A (Duration 1-12 weeks):

Participants will be given Vitamin D (VD) supplementation at a dose of 600,000 IU along with Calcium 1000 mg/day.

Mid-Point (At 12 weeks):

Patients will have a consultation for clinical interpretation. They will undergo biochemical assessment, including the estimation of Insulin Resistance, Free Androgen Index, and Total Antioxidant Capacity.

After 12 weeks They will receive standard treatment for Polycystic Ovary Syndrome (PCOS), which includes Glucophage XR 750 mg once at dinner for 15 days, then twice daily. Capsule Progeffik 100 mg once at night every 3 weeks, then 1 week off and Calcium 1000 mg/day

Intervention Details for Group B (Duration 1-12 weeks):

Participants in Group B will receive standard PCOS treatment mentioned earlier:

Glucophage XR 750 mg once at dinner for 15 days, then twice daily. Capsule Progeffik 100 mg once at night every 3 weeks, then 1 week off. Additionally, they receive Calcium 1000 mg/day.

Mid-Point (At 12 weeks):

Patients will have a consultation for clinical interpretation. They will undergo biochemical assessment, including the estimation of Insulin Resistance, Free Androgen Index, and Total Antioxidant Capacity.

Intervention Details for Group A (After 12 weeks)

They will receive VD supplementation (600,000 IU) during this time and continue to receive Calcium 1000 mg/day.

Calculations of HOMA-IR and Free Androgen Index will be done at 12 and 24 weeks and the results will be compared.

{HOMA-IR: HOMA- IR index, a commonly used marker of IR, will be calculated using the formula: HOMA-IR = fasting glucose levels [mmol/L] × fasting insulin levels [μU/mL]/22.5 Free Androgen Index will be derived from TT and SHBG, normally measured in nanomoles per liter. FAI =100 (TT /SHBG)}

ELIGIBILITY:
Inclusion Criteria:

* Recently diagnosed PCOS with presence of at least 2 of these 3 elements: clinical or biochemical signs of hyperandrogenism, chronic anovulation and polycystic ovaries (1) (from reports of available routine TVS), with VDD serum levels VD <20 ng/ml(10), age range 18- 45 years, from all ethnic background will be included.

Exclusion Criteria:

* : Exclusion of subjects will be done by the Co-Principal Investigators (Co-PI) after history, examination and complete evaluation in the respective clinics. All female subjects meeting any of the following criteria will be excluded from the study

  * Pregnancy
  * Hypercalcemia (plasma calcium concentrations> 2.65 mmol/L)
  * Tuberculosis or other granulomatous disorders
  * Chronic liver disease or alanine transaminase (ALT) level 3 times higher than the normal limit, chronic
  * Kidney disease or serum creatinine >2.0 mg/dL,
  * Drug Therapies: VD replacement ; participants who had received VD injection in the last 3 months prior to recruitment in the study, oral contraceptives, hormonal replacement therapy, glucocorticoids, calcium supplementation, insulin-sensitizing drugs (incretin mimetic drugs, thiazolidinedione, sulfonylurea), lipid-lowering drugs or other drugs affecting insulin sensitivity or serum androgens (e.g., niacin, corticosteroids, beta-blockers, calcium channel blockers, thiazide diuretics), anti-epileptics, anti-retroviral, cholestyramine, anti-fungal, statins, H2 blockers, immunosuppressant, chemotherapeutic agents, antimicrobials (Rifampicin, Isoniazid, Hydroxychloroquine) or any other drug modifying lipid metabolism in the previous 3 months prior to study
  * Suffering from congenital adrenal hyperplasia, Cushing's syndrome, androgen-secreting tumors, type 2 Diabetes Mellitus, renal, hepatic or thyroid disorders, hyperparathyroidism, malabsorption syndromes, Chronic Kidney Disease, Hepatic failure, cystic fibrosis, vaginal bleeding of unknown etiology or /and suffering from COVID-19 (within 3 months).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 142 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
hyperandrogenism | 24 weeks
  hyperandrogenism by Free Androgen Index [Total Testosterone, Steroid Hormone Binding Globulin
insulin Resistance | 24 weeks
  HOMA-IR (serum Insulin, Fasting Blood Glucose)
oxidative stress | 24 weeks
  Total Antioxidant Capacity

CONTACTS AND LOCATIONS:
Overall Officials: Rehana Rehman, PhD, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/51/NCT06045351/Prot_001.pdf